CLINICAL TRIAL: NCT06288711
Title: Novel Telemedicine-Delivered Prolonged Exposure Therapy for Treating PTSD in Individuals With OUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Peck, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRBSS #STUDY00002538; R01DA057308 (NIH)
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Posttraumatic Stress Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as usual (TAU) (Active Comparator): Participants randomized to TAU will continue to receive standard buprenorphine or methadone maintenance treatment from their current treatment provider and complete follow-up assessments as described above. However, they will not receive posttraumatic stress disorder treatment. Staff will mail participants an emergency naloxone kit containing two naloxone doses with simple instructions, a list of resources and contact information for mental health providers and other relevant resources in their community and assistance contacting any resources of interest.
  Interventions: Behavioral: Treatment as usual
- Prolonged exposure therapy (PE) (Experimental): In addition to receiving standard buprenorphine- or methadone-maintenance treatment from their current provider and completing scheduled assessments as described above, PE participants will also receive 12 individual sessions of prolonged exposure therapy scheduled weekly over the 12-week treatment period and delivered via a secure and university-supported telemedicine platform. Beginning in study week 1, PE participants will complete weekly 60-minute telemedicine-delivered prolonged exposure therapy sessions provided by doctoral or master's level therapists trained in prolonged exposure therapy.
  Interventions: Behavioral: Prolonged exposure therapy; Behavioral: Treatment as usual
- Prolonged exposure therapy + attendance contingent financial incentives (PE+) (Experimental): Participants assigned to the PE+ condition will receive the procedures noted above for the PE group plus financial incentives delivered contingent upon completion of PE sessions.
  Interventions: Behavioral: Prolonged exposure therapy; Behavioral: Financial incentives; Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Prolonged exposure therapy — Twelve weekly 60-minute telemedicine-delivered prolonged exposure therapy sessions provided by therapists trained in prolonged exposure therapy.
  Arms: Prolonged exposure therapy (PE); Prolonged exposure therapy + attendance contingent financial incentives (PE+)
Behavioral: Financial incentives — Financial incentives contingent upon completion of prolonged exposure therapy sessions
  Arms: Prolonged exposure therapy + attendance contingent financial incentives (PE+)
Behavioral: Treatment as usual — Continued standard buprenorphine or methadone maintenance treatment from current treatment provider.

SUMMARY:
Among individuals with opioid use disorder (OUD), posttraumatic stress disorder (PTSD) presents a significant clinical challenge. The prevalence of PTSD is substantially higher in individuals with OUD than in the general population, with nearly 90% reporting lifetime trauma exposure and 33% meeting diagnostic criteria for PTSD. The primary objective of this study is to evaluate the efficacy of a novel telemedicine-delivered prolonged exposure therapy protocol for improving PE attendance and reducing PTSD symptom severity in individuals with concurrent PTSD and OUD.

DETAILED DESCRIPTION:
Nearly 90% of individuals with opioid use disorder (OUD) report lifetime trauma exposure and 33% meet criteria for posttraumatic stress disorder (PTSD). Patients with co-occurring PTSD and OUD are at significantly greater risk for poor substance use and mental health outcomes vs. those with OUD alone. Although Prolonged Exposure (PE) therapy is a first-line treatment for PTSD, its efficacy is commonly undermined by poor attendance.

The primary objective of this study is to evaluate the efficacy of a novel telemedicine-delivered prolonged exposure therapy protocol for improving PE attendance and reducing PTSD symptom severity in individuals with concurrent PTSD and OUD. In this randomized trial, adults with PTSD (N = 135) who are currently maintained on MOUD will be randomly assigned to one of three conditions: (a) Treatment as usual (TAU), (b) Prolonged exposure therapy (PE), or (c) Prolonged exposure therapy + attendance-contingent financial incentives (PE+). Participants randomized to the TAU condition will continue to receive standard MOUD treatment from their current treatment provider and complete remotely-administered assessments of PTSD symptoms, psychosocial functioning and drug use with an evaluator trained in the administration of all study measures and blinded to treatment condition at intake, monthly during the 12-week intervention, and at 3- and 6-months post-study, but will not receive PTSD treatment. In addition to receiving continued MOUD treatment from their current provider and completing assessments as above, participants assigned to PE will also receive telemedicine-delivered PE consisting of 12 weekly, individual sessions with trained master's- or doctoral-level therapists. PE sessions consist of imaginal exposure (i.e., revisiting and recounting traumatic memories) and processing the memory (i.e., discussing thoughts and feelings related to revisiting the memory). Participants also complete homework assignments consisting of repeated listening to a recording of the imaginal exposure and repeated in vivo exposure to safe situations that have previously avoided because of trauma-related distress. Participants assigned to the PE+ condition will receive the procedures noted above for the PE condition plus attendance-contingent financial incentives delivered immediately following completion of telemedicine-delivered PE sessions via a digital payment delivery platform.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Maintained on a stable methadone or buprenorphine dose for >1 month prior to the study
* Meet current DSM-5 posttraumatic stress disorder criteria based on the Clinician Administered PTSD Scale for DSM-5
* Participants receiving psychotropic medications must be maintained on a stable dose for >1 month prior to enrollment.

Exclusion Criteria:

* Current delusions or hallucinations, unstable bipolar disorder, imminent risk for suicide as assessed by the Mini International Neuropsychiatric Interview
* Cognitive impairment as evidenced by scores <22 on the Videoconference-based Mini Mental Status Examination (MMSE; Folstein, et al., 1975)
* Enrolled in another ongoing evidence-based treatment for PTSD.
* Pregnancy as verified by pregnancy test
* No access to cellular service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Prolonged exposure therapy session attendance | From baseline to week 12
  Percentage of scheduled prolonged exposure therapy sessions attended
Prolonged exposure therapy completion | From baseline to week 12
  Percentage of participants completing eight or more prolonged exposure therapy sessions
Change in posttraumatic stress disorder symptom severity - clinician rated | From baseline to week 12
  Change in posttraumatic stress disorder symptom severity as measured by Clinician Administered PTSD Scale (CAPS-5) for clinician-rated posttraumatic stress symptoms. The CAPS-5 is a 30-item structured interview. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 PTSD symptoms, each with severity scores ranging from 0-4. The overall total severity score for CAPS-5 ranges from 0-80, with lower scores representing better outcomes (less severe PTSD).

SECONDARY OUTCOMES:
Change in non-prescribed drug use - objective | From baseline to week 12 and 3, 6 months post-study
  Change in non-prescribed drug use will be measured by the overall percentage of urine drug screens verified to be positive for non-prescribed opioids (e.g., heroin, methadone, buprenorphine, oxycodone, fentanyl) and non-opioid drugs (e.g., cocaine, amphetamines, benzodiazepines) during the treatment period.
Change in non-prescribed drug use - self-reported | From baseline to week 12 and 3, 6 months post-study
  Time Line Follow Back (TLFB) to measure non-prescribed drug use.
Change in opioid craving | From baseline to week 12
  Single item measure (range: 0-100) of craving for opioids.
Medications for opioid use disorder treatment retention | From baseline to week 12 and 3, 6 months post-study
  Percentage of participants retained in medications for opioid use disorder treatment
Prolonged exposure therapy acceptability | From baseline to week 12
  Treatment Acceptability/Adherence Scale to measure treatment acceptability
Satisfaction with prolonged exposure therapy delivered via telemedicine | From baseline to week 12
  Telemedicine Satisfaction Questionnaire to measure satisfaction with treatment delivered via telemedicine
Prolonged exposure therapy homework adherence | From baseline to week 12
  Homework adherence questionnaire to measure prolonged exposure therapy homework adherence
Change in posttraumatic stress disorder symptom severity - self-reported | From baseline to week 12
  Change in posttraumatic stress disorder symptom severity as measured by PTSD Checklist for DSM-5 (PCL-5) for self-reported posttraumatic stress symptoms. The PCL-5 is a 20-item self-report measure that assesses the 20 symptoms of PTSD. The rating scale is 0-4 for each symptom/item, and overall scores range from 0-80, with lower scores representing better outcomes (less severe PTSD).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vemont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No